CLINICAL TRIAL: NCT03540888
Title: Effect of Deep Transverse Friction Massage Versus Stretching Techniques on Performance Among Lebanese and Syrian Football Players
Brief Title: Effects of Deep Friction Vs Stretching Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Ali FAKHRO, DPT (Other)
Responsible Party: Sponsor-Investigator, Mohammed Ali FAKHRO, DPT, Coordinator, Lebanese German University
Organization: Lebanese German University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Deep transverse friction
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Deep Transverse Friction Massage
Keywords: Dynamic Stretching; Static Stretching; Manual Therapy

STUDY DESIGN:
Intervention Model Description: In order to compare the effects of DTFM to static and dynamic stretching techniques, participants were randomly assigned to one of three groups (a) DTFM group, (b) Dynamic stretching group, and (c) Static stretching group, and were followed- up over four weeks period.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Transverse Friction Massage group (Experimental): Deep transverse friction massage group. Participants were taught by one of the examiners how to sit and perform pre-exercise self-massages on their tested leg musculotendinous junction (MTJ). The procedure consisted of applying friction massage by fingertips transversely to the hamstrings tendon, in a sitting position. The tendon was located over four finger widths proximal to the medial and lateral epicondyles of the femur. One examiner carefully monitored how the technique was performed to assure the precision of the application. This massage technique was applied over a duration of 30 seconds.
  Interventions: Other: Deep transverse Friction Massage
- Dynamic stretching intervention (Active Comparator): The dynamic stretching intervention was included for its positive effects on agility and muscle strength. Participants in this group, swung their tested leg actively into hip flexion while keeping their knee fully extended and their ankle fully plantar flexed until a stretch was felt in the posterior thigh. This was repeated over 30 seconds and included in the participant's warm-up phase.
  Interventions: Other: Dynamic stretching intervention
- Static stretching intervention (Active Comparator): In the static stretching intervention, all participants laid on the floor in a supine position with both feet pointing upwards, with the tested limb in full knee extension and the foot in a relaxed position. The tested limb was moved up passively to a point of slight pain or discomfort at the posterior aspect of the thigh. This technique puts the hamstrings muscle at its greatest possible length. This position should be held for 30 seconds and was performed three times for a total of one minute and 30 seconds, 15 minutes after a match or training. The contralateral leg was stabilized by means of another collaborator in order to prevent compensation by rotation or elevation of the pelvis.
  Interventions: Other: Static stretching intervention

INTERVENTIONS:
Other: Deep transverse Friction Massage — The procedure consisted of applying friction massage by fingertips transversely to the hamstrings tendon, in a sitting position. The tendon was located over four finger widths proximal to the medial and lateral epicondyles of the femur
  Other Names: DTFM
  Arms: Deep Transverse Friction Massage group
Other: Dynamic stretching intervention — Participants in this group, swung their tested leg actively into hip flexion while keeping their knee fully extended and their ankle fully plantar flexed until a stretch was felt in the posterior thigh. This was repeated over 30 seconds and included in the participant's warm-up phase.
  Arms: Dynamic stretching intervention
Other: Static stretching intervention — In the static stretching intervention, all participants laid on the floor in a supine position with both feet pointing upwards, with the tested limb in full knee extension and the foot in a relaxed position. The tested limb was moved up passively to a point of slight pain or discomfort at the posterior aspect of the thigh. This technique puts the hamstrings muscle at its greatest possible length. This position should be held for 30 seconds and was performed three times for a total of one minute and 30 seconds, 15 minutes after a match or training. The contralateral leg was stabilized by means of another collaborator in order to prevent compensation by rotation or elevation of the pelvis.
  Arms: Static stretching intervention

SUMMARY:
Flexibility, agility and muscle strength are key factors to either win or lose a game. Recently the effect of a new technique, deep transverse friction massage (DTFM), on muscle extensibility, strength and agility and injury occurrence has been examined, as compared to traditional stretching techniques.

DETAILED DESCRIPTION:
Background: Flexibility, agility and muscle strength are key factors to either win or lose a game. Recently the effect of a new technique, deep transverse friction massage (DTFM), on muscle extensibility, strength and agility and injury occurrence has been examined, as compared to traditional stretching techniques.

Hypothesis/Purpose: To compare the effect of DTFM vs static and dynamic stretching techniques on hamstrings extensibility, agility and strength among Lebanese and Syrian football players.

Study Design: This study is a single-blinded prospective longitudinal randomized control trial (RCT).

Methods: Football players were randomized into three intervention groups. Straight leg raise (SLR), T-drill, and 1 repetition maximum (RM) tests were used to measure extensibility, agility and maximal muscle strength respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Football player
* Physically active (1 to 3 hours of football per week).

Exclusion Criteria:

• Under the age of 18 and over 35 years who presented with an injury to the musculoskeletal system.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in flexibility was measured by Straight leg raise test. | baseline, on the first session; (2) 15 minutes, after the first intervention (acute phase); and (3) after four weeks
  Straight leg raise (SLR) is a widely used outcome measure used to assess the extensibility of the hamstrings muscle. SLR was first applied to all participants across the groups. All football players laid supine and taught to relax during testing. The tested limb was raised by a volunteer therapist with the knee in full extension and the foot in a relaxed position. The other lower limb was stabilized in a neutral hip rotation and full knee extension by another volunteer. The test was stopped once the therapist felt a strong resistance, or when the pelvic rotation was noted. Then, the assessor placed the goniometer over the greater trochanter, with one arm aligning the lateral femoral condyle, and the other arm aligning parallel to the ground, in a direction to the mid-axillary line and recorded the hip angle. The scores were recorded as degrees of range of movement.
Change in agility was measured by T-Drill test. | baseline, on the first session; (2) 15 minutes, after the first intervention (acute phase); and (3) after four weeks
  The T-Drill has been proven to be a highly reliable testing measurement. Footballers were instructed on how to perform the T-Drill and on the test procedures. Then, they were instructed to jog for 2 min to warm-up. The participants performed the T-drill twice and the trial with the best time was taken for analysis by the mean of an alert assessor with a stopwatch. Results were measured in seconds and scores were interpreted as (1) excellent, < 9.5; (2) good, 9.5-10.5; (3) average, 10.5-11.5; and (4) poor, > 11.5.
Change in Strength was measured by one repetition maximum (1RM) tests | baseline, on the first session; (2) 15 minutes, after the first intervention (acute phase); and (3) after four weeks
  After a rest time of 5 min, participants were guided to the knee flexors strengthening machine (hamstrings curl machine) for one repetition maximum (1RM) testing. Resistance was placed just proximal to the posterior part of the calcaneus bone. Footballers performed first specific warm-up, consisting of a set of ten repetitions of knee flexion, with a light load. Afterwards, for safety reasons, an estimation of hamstring 1RM was calculated using Brzycki formula [Weight lifted ÷ (1.0278 - (0.0278 × Number of repetitions)]. This formula exhibited a relatively low level of bias (1.6 to 0 kg). Maximal voluntary strength was recorded in kilograms.

SECONDARY OUTCOMES:
Change in injury occurrence rate | baseline, after 4 weeks.
  Measured by recording if any injury affected the players.

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese German University, Jounieh, Keserwan, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03540888/Prot_SAP_002.pdf